CLINICAL TRIAL: NCT01846624
Title: A Phase 2 Study of Decitabine in Combination With Midostaurin (PKC412) for Elderly Patients With Newly Diagnosed FLT3-ITD/TKD Positive Acute Myeloid Leukemia
Brief Title: Decitabine and Midostaurin in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual factor
Sponsor: David Iberri (Other)
Responsible Party: Sponsor-Investigator, David Iberri, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25737; HEMAML0022 (Registry Identifier: OnCore)
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2018-09-07 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Acute Myeloid Leukemia (AML) With Multilineage Dysplasia Following Myelodysplastic Syndrome, in Adults; AML (Adult) With 11q23 (MLL) Abnormalities; AML (Adult) With Del (5q); AML (Adult) With Inv (16) (p13; q22); AML (Adult) With t (16;16) (p13; q22); AML (Adult) With t (8; 21) (q22; q22); Secondary AML (Adult); Untreated AML (Adult)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Decitabine; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine, then midostaurin (Experimental): INDUCTION THERAPY Subjects receive decitabine intravenously (IV) over 1 hour on days 1 to 10 and midostaurin orally (PO) twice daily (BID) on days 11 to 28. Treatment repeats every 28 days until documented bone marrow response is achieved or for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients achieving documented bone marrow response by course 6 continue treatment with induction therapy; patients achieving response after course 6 proceed to post-remission therapy.
  POST-REMISSION THERAPY Subjects receive decitabine IV over 1 hour on days 1 to 5 and midostaurin PO BID on days 6 to 28. Treatment repeats every 28 days for up to 12 courses (including induction therapy) in the absence of disease progression or unacceptable toxicity.
  After completion of study treatment, patients are followed up for up to 1 year.
  Interventions: Drug: Decitabine; Drug: Midostaurin

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC; Dacogen
Drug: Midostaurin — Given PO
  Other Names: N-benzoyl-staurosporine; PKC412

SUMMARY:
This phase 2 study evaluates the sequential combination of decitabine then midostaurin for the treatment of newly-diagnosed acute myeloid leukemia (AML) in older patients.

DETAILED DESCRIPTION:
Treatment with decitabine, a cytidine analog, then midostaurin, a multi-target protein kinase inhibitor (PKI), may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed acute myeloid leukemia (AML) per the World Health Organization [WHO] 2008 classification [except t (15; 17)], including:

  * De novo AML
  * Secondary AML
  * Secondary AML arising from previously-diagnosed myelodysplastic syndromes (MDS) treated with deoxyribonucleic acid (DNA) methyltransferase inhibitor (DNMTi) (ie, decitabine or azacitidine)
* FLT3-ITD mutation confirmed in bone marrow aspirate
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN)
* Serum bilirubin ≤ 2.5 ULN
* Serum creatinine ≤ 1.5 mg/dL and/or creatinine clearance ≥ 50 mL/min
* Ejection fraction ≥ 50% by echocardiogram
* Unwillingness or inability to receive conventional chemotherapy
* Ability to understand and the willingness to sign a written informed consent document
* Ability to adhere to the study visit schedule and other protocol requirements
* Life expectancy > 2 months

Exclusion Criteria:

* Receiving concomitant treatment with other anti-neoplastic agents (EXCEPTION: hydroxyurea). Prior treatment with DNMTi therapy (ie, decitabine or azacitidine) for MDS is allowed
* Received anti-neoplastic treatment within 4 weeks prior to enrollment (EXCEPTION: hydroxyurea)
* Received any surgical procedure, excluding central venous catheter placement or other minor procedures (eg, skin biopsy) within 14 days of study day 1
* Received any investigational agent within 4 weeks prior to enrollment
* Previous or current history of a myeloproliferative disease
* Known active central nervous system (CNS) malignancy
* Any other known disease (except carcinoma in-situ), concurrent severe and/or uncontrolled medical condition which could compromise participation in the study (eg, uncontrolled diabetes; cardiovascular disease including congestive heart failure; myocardial infarction within 6 months with poorly controlled hypertension; chronic renal disease; active uncontrolled infection)
* Active opportunistic infection or treatment for opportunistic infection within 4 weeks of first day of study drug dosing
* Known confirmed diagnosis of human immunodeficiency virus (HIV) infection or active viral hepatitis
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of midostaurin
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to midostaurin and/or decitabine
* Impaired cardiac function including any of the following:

  * Screening electrocardiogram (ECG) with a corrected QT interval (QTc) > 450 msec
  * Bradycardia defined as heart rate (HR) < 50 beats per minute (bpm)
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Patients with myocardial infarction or unstable angina < 3 months prior to starting study drug
  * Congestive heart failure (CHF) New York (NY) Heart Association class 3 or 4
* Inability to swallow or absorb drug
* Other medical or psychiatric illness or organ dysfunction or laboratory abnormality which in the opinion of the investigator would compromise the patient's safety or interfere with data interpretation
* Unwillingness or inability to comply with the protocol
* Pregnant
* nursing (lactating)
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are using highly effective methods of contraception during dosing and for 3 months after midostaurin medication; highly effective contraception methods as follows:

  * Total abstinence, when this is in line with the preferred and usual lifestyle of the subject [periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception]
  * Female sterilization (surgical bilateral oophorectomy with or without hysterectomy; or tubal ligation at least six weeks before taking study treatment). In case of oophorectomy alone, reproductive status must be confirmed by follow-up hormone level assessment
  * Male sterilization, at least 6 months prior to screening (for female subjects on the study, the vasectomized male partner should be the sole partner for that subject)
  * Combination of any two of the following (a+b or a+c, or b+c):

    * Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), eg, hormone vaginal ring or transdermal hormone contraception. For oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07-22 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Iberri, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Dohner H, Estey EH, Amadori S, Appelbaum FR, Buchner T, Burnett AK, Dombret H, Fenaux P, Grimwade D, Larson RA, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz MA, Sierra J, Tallman MS, Lowenberg B, Bloomfield CD; European LeukemiaNet. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood. 2010 Jan 21;115(3):453-74. doi: 10.1182/blood-2009-07-235358. Epub 2009 Oct 30. PMID 19880497

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine, Then Midostaurin: INDUCTION THERAPY Subjects receive decitabine intravenously (IV) over 1 hour on days 1 to 10 and midostaurin orally (PO) twice daily (BID) on days 11 to 28. Treatment repeats every 28 days until documented bone marrow response is achieved or for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients achieving documented bone marrow response by course 6 continue treatment with induction therapy; patients achieving response after course 6 proceed to post-remission therapy.
  POST-REMISSION THERAPY Subjects receive decitabine IV over 1 hour on days 1 to 5 and midostaurin PO BID on days 6 to 28. Treatment repeats every 28 days for up to 12 courses (including induction therapy) in the absence of disease progression or unacceptable toxicity.
  After completion of study treatment, patients are followed up for up to 1 year.
  Decitabine: Given IV
  Midostaurin: Given PO
Period: Overall Study
Arm/Group | Decitabine, Then Midostaurin
Started | 13
Completed | 12
Not Completed | 1
Not completed — Died during induction, no midostaurin | 1

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine, Then Midostaurin
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate
Description: The complete remission (CR) rate, or complete response rate, is reported as the sum and proportion of participants that achieved CR or CR with incomplete blood count recovery (CRi), within 12 months of starting midostaurin treatment.
  * Complete remission (CR): Bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) > 1000/μL; platelet count > 100,000/μL; independence of red cell transfusions.
  * CR with incomplete recovery (CRi): All CR criteria except for ANC < 1000/μL or platelet count < 100,000/μL.
  * Partial remission (PR): All hematologic criteria of CR; except decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Time Frame: Up to 1 year
Population: Only participants that started midostaurin therapy are included in the complete response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine, Then Midostaurin
Number analyzed (Participants) | 12
Participants | 8

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response rate (ORR) was assessed as the number and proportion of participants who received midostaurin and achieved a partial response (PR), complete response (CR), or complete response with incomplete blood count recovery (CRi).
  * Complete remission (CR): Bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) > 1000/μL; platelet count > 100,000/μL; independence of red cell transfusions.
  * CR with incomplete recovery (CRi): All CR criteria except for ANC < 1000/μL or platelet count < 100,000/μL.
  * Partial remission (PR): All hematologic criteria of CR; except decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Time Frame: up to 1 year
Population: Only participants that started midostaurin therapy are included in the response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine, Then Midostaurin
Number analyzed (Participants) | 12
Participants | 10

3. Secondary Outcome: Median Duration of Response (DoR)
Description: Response was assessed by evaluations conducted every 3 cycles (12 weeks). Once documented as partial response (PR), complete response (CR), or complete response with incomplete blood count recover (CRi), response status was confirmed every 12 weeks. In responding participants, duration of response was assessed from the start of treatment through the last documented response before documented progressive disease or death. The outcome is reported as the median value for duration of response, with full range.
  * CR: Bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; ANC > 1000/μL; platelet > 100,000/μL; independence of red cell transfusions.
  * CRi: All CR criteria except ANC < 1000/μL or platelet count < 100,000/μL.
  * PR: All hematologic criteria of CR; except decrease of bone marrow blast percentage to 5% to 25%; & decrease of pretreatment bone marrow blast percentage by at least 50%.
Time Frame: Up to 1 year
Population: Does not include participants who did not achieve a documented clinical response. Participants who withdrew to receive hematopoietic cell transplant (HCT) are censored at the last assessment of response prior to HCT.
Measure: Median (Full Range); unit: weeks
Arm/Group | Decitabine, Then Midostaurin
Number analyzed (Participants) | 10
weeks | 24 [12 to 36]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is reported as the number and proportion of participants who did not receive hematopoietic cell transplantation, and who did not experience disease progression or death for any reason within 2 years after starting midostaurin treatment.
  Progressive disease: Bone marrow blasts ≥ 5%; or reappearance of blasts in the blood; or development of extramedullary disease.
Time Frame: Up to 2 years
Population: Only participants that started midostaurin therapy, and did not withdraw for hematopoietic cell transplantation, are included in the progression-free survival assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine, Then Midostaurin
Number analyzed (Participants) | 9
Participants | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Survival is reported as the number and proportion of participants that received midostaurin who remained alive 2 years after starting midostaurin treatment.
Time Frame: Up to 2 years
Population: Only participants that started midostaurin therapy are included in the overall survival assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Decitabine, Then Midostaurin
Number analyzed (Participants) | 12
Participants | 2

ADVERSE EVENTS:
Arm/Group | Decitabine, Then Midostaurin
All-Cause Mortality (participants affected / at risk) | 11/13
Serious Adverse Events (participants affected / at risk) | 13/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine, Then Midostaurin (N=13)
Renal failure (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Hematoma, subdural (Nervous system disorders) | 1 (1)
Unresponsive (Nervous system disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) — Vision loss in right eye
Pain, eye (Eye disorders) | 1 (1) — Right eye
Kidney stones (nephrolithiasis) (General disorders) | 1 (1) — Right kidney
Swelling in arms and legs (peripheral edema) (General disorders) | 1 (1)
Bowel obstruction (Gastrointestinal disorders) | 1 (1) — Partial
Bleeding (hemmorhage) (Gastrointestinal disorders) | 1 (1)
Neutropenic fever (Immune system disorders) | 13 (24)
Tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) — 1 event was fatal
Herpetic stomatitis (Infections and infestations) | 1 (1) — Herpes simplex virus (HSV)
Sepsis (Infections and infestations) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Anoxic brain injury (Respiratory, thoracic and mediastinal disorders) | 3 (3) — 1 event was fatal
Shortness of breath (dyspnea) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Low oxygen in blood (hypoxemia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Low oxygen in tissues (hypoxia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Excess fluid around the lungs (pleural effusion) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Includes 1 instance of bilateral pneumonia
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 (4) — 2 events fatal
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decitabine, Then Midostaurin (N=13)
Arrhythmia (Cardiac disorders) | 5 (5) — Electrocardiogram abnormality
Hypertension (Cardiac disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hearing loss (Nervous system disorders) | 1 (1)
Altered mental status (Nervous system disorders) | 2 (2)
Confusion (Nervous system disorders) | 1 (1)
Agitation (Nervous system disorders) | 1 (1)
Delirium (Nervous system disorders) | 1 (1) — Sundowning
Lighted-headed (Nervous system disorders) | 1 (1)
Tinnitus (Nervous system disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1) — Dizziness
Sleep disorders (Nervous system disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Distress (Nervous system disorders) | 1 (1)
Memory loss (Nervous system disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1) — Photophobia and blurred vision
Nausea (Gastrointestinal disorders) | 3 (3)
Taste alteration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Abdominal / epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Cough (Gastrointestinal disorders) | 5 (5)
Abdominal pain with bloating (Gastrointestinal disorders) | 2 (2)
Poor appetite (Gastrointestinal disorders) | 2 (2)
Metallic taste (Gastrointestinal disorders) | 1 (1)
Stomatitis (Infections and infestations) | 4 (4) — Herpes simplex virus
Cellulitis (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Limb edema (General disorders) | 5 (5)
Weight loss (General disorders) | 4 (4)
Alopecia (General disorders) | 3 (3)
Dysgeusia (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Mouth sores (General disorders) | 2 (2)
Fall (General disorders) | 1 (1)
Fracture (General disorders) | 1 (1) — Left lower leg
Tingling and weakness (General disorders) | 1 (1) — Lower extremities
Foot drop (General disorders) | 1 (1)
Blood-tinged sputum (General disorders) | 1 (1)
Pain on right thumb (General disorders) | 1 (1)
Shoulder pain (General disorders) | 2 (2)
Facial flushing (General disorders) | 1 (1)
Multi-organ dysfunction (General disorders) | 1 (1)
Leg pain (General disorders) | 1 (1)
Worsening of neuropathy (General disorders) | 1 (1) — In the extremities
Pain on left side of tongue (General disorders) | 1 (1)
Neck pain (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 3 (3)
Desquamation on extremities (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Lip lesions (Skin and subcutaneous tissue disorders) | 2 (2)
Lesion in buccal mucosa (Skin and subcutaneous tissue disorders) | 3 (3) — Oral thrush
Diaphoretic (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Viral illness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased lung breathing sounds (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Invasive lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neutropenic fever (Blood and lymphatic system disorders) | 4 (4)
Hemoptysis (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 5 (5)
Chills (Blood and lymphatic system disorders) | 1 (1)
Disease Progression (Blood and lymphatic system disorders) | 4 (4) — Acute myeloid leukemia
Lymphocytopenia (Blood and lymphatic system disorders) | 1 (1)
Increased transfusions (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1)
Cytopenia (Blood and lymphatic system disorders) | 1 (1)
Transfusion reaction to platelets (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Restless legs (Metabolism and nutrition disorders) | 1 (1)
Acute renal failure (Metabolism and nutrition disorders) | 3 (3)
Aspartate aminotransferase elevated (Metabolism and nutrition disorders) | 1 (1)
Alanine aminotransferase elevated (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No